CLINICAL TRIAL: NCT06232577
Title: 5x-Multiplier vs 3-Tier Model for Discharge Opioid Prescriptions After Intra-abdominal Cancer Surgery: A Randomized Clinical Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0818; NCI-2024-00632 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Intra-abdominal Cancer
MeSH Terms: interventions — Hydrocodone; Tramadol; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5x-Multiplier Model (Experimental): In this group, you will be given 5 times the amount of opioid medication you needed on your last day in the hospital. You would then use this supply plus standard non-narcotic pain medications.
  Interventions: Drug: Hydrocodone; Drug: Tramadol; Drug: Oxycodone
- 3-Tier Model (Experimental): The total amount of opioid medication you needed on your last day in the hospital to set a maximum number of opioid medications at discharge (up to 30).
  Interventions: Drug: Hydrocodone; Drug: Tramadol; Drug: Oxycodone

INTERVENTIONS:
Drug: Hydrocodone — Given by PO
Drug: Tramadol — Given by PO
Drug: Oxycodone — Given by PO
  Other Names: ETH-Oxydose™ [DSC]; OxyContin®; OxyIR®; Roxicodone®

SUMMARY:
To compare 2 different models for prescribing opioid pain medication to provide better pain control to participants with an abdominal cancer who are having surgery.

DETAILED DESCRIPTION:
Primary Objectives:

The co-primary objectives of this study are as follows:

1. To determine differences in the initial OME prescribed upon discharge between each algorithm/model.

1. To determine OME usage by day 14 after hospital discharge.

Secondary Objectives:

Secondary objectives are as follows:

1. To determine rates of patients with zero OME upon discharge.
2. To determine rates of OME refill requests and completions at 15- and 30-days post-operation.
3. To determine number of unused or leftover pills at 15- and 30-days post- operation
4. To determine persistent opioid use at 30-days, 3-months, and 6-months post-operation
5. To elucidate patient, prescriber, and oncologic factors predictive of persistent opioid use
6. To assess quality of life using patient-reported outcomes at 30-days, 3-months, and 6-months post-operation.
7. To determine patient satisfaction with either prescribing model.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age
* Participants undergoing any of the following abdominal surgeries on an elective basis at MD Anderson Cancer Center:
* Open pancreatectomy
* Open hepatectomy
* Open resection of retroperitoneal sarcoma
* Open nephrectomy
* Open cytoreductive surgery (in ovarian cancer)
* Participants with a planned inpatient admission of at least 48 hours after surgery
* Opioid-naive patients who use less than or equal to 7.5 mg OME per day (on average) during the 30 days prior to consent
* Participants able to understand and willing to sign an informed consent document
* English and non-English-speaking participants

Exclusion Criteria:

* Participants requiring non-elective (emergent or urgent) surgery will be excluded
* Participants with a current or previous history of substance abuse disorder, including alcohol or drugs
* Participants prescribed long-acting chronic pain medications
* Participants using hydromorphone or fentanyl or under the care of a chronic pain specialist
* Participants unable or unwilling to participate in follow-up study requirements (e.g., QOL surveys, opioid log)
* Participants discharged on palliative or hospice care
* Participants with a history of allergic reactions to opioids
* Participants enrolled in any other opioid discharge protocol
* Participants who are pregnant
* Participants who are cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Wei D Tzeng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Fields BC, Newhook TE, Lillemoe HA, Qiao W, Karam JA, Matin SF, Meyer LA, Tzeng CD. 5x-Multiplier vs 3-Tier Model for Discharge Opioid Prescriptions After Intra-Abdominal Cancer Surgery: Randomized Clinical Trial Protocol. Adv Cancer Educ Qual Improv. 2025;1(1):19. doi: 10.52519/aceqi.25.1.1.a19. PMID 40583965
- See also: MD Anderson Cancer Center — http://www.mdanderson.org